CLINICAL TRIAL: NCT07143643
Title: The Effect of Using Escape Room Method on Nursing Studentsˈ Self-Efficacy, Team Collaboration and Anxiety in Nursing Process Teaching
Brief Title: The Effect of Escape Room Method in Nursing Process Teaching
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Yasemin Kıyak Yorulmaz, Principal Investigator Phd candidate of nursing, Bezmialem Vakif University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: YKİYAK
Record Dates: First submitted 2025-08-20; First posted 2025-08-27 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-08

CONDITIONS: Nursing Education; ESCAPE ROOM; Nursing Students
Keywords: Escape Room Method; Self-Efficacy; Team Collaboration; Nursing process; Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Participant Group (Experimental): Experimental: Escape room simulation group- Within the scope of the theoretical training on the nursing process, a two-week education will be provided. Afterwards, the students in this group will be divided into five groups of seven students each and will participate in an escape room game based on a case prepared regarding the nursing process.
  Interventions: Other: Excape room game
- Control group (No Intervention): Control group: Within the scope of the theoretical training on the nursing process, a two-week education will be provided. Afterwards, using the traditional teaching method, five groups of seven students each will examine the same case scenario applied to the experimental group within the framework of the nursing process for 60 minutes. The groups will work independently of each other in the same classroom environment and, together with the researcher, will analyze the case within the framework of the nursing process for 60 minutes using traditional teaching methods such as question-and-answer and discussion.

INTERVENTIONS:
Other: Excape room game — Application of Research:The escape room game scenario prepared by the researchers was designed according to the steps of the Nursing Process. The game consists of five stages, each conducted at different stations, and each stage includes various clues and activities. The stages were organized to cover the steps of the Nursing Process: "Assessment, Nursing Diagnosis, Planning, Implementation, and Evaluation." Before starting the game, the students who will participate will be informed about the expected objectives, the game rules, and the duration. In addition, it will be stated that each group must select a group leader. The students will be given a total of 60 minutes to answer the questions in each stage, assemble puzzle pieces, unlock locked boxes, follow the clues, and find the exit key in order to leave the room. The students will be expected to complete the tasks at the stations prepared in accordance with the Nursing Process stages and to exit the room within the allotted time.
  Arms: Participant Group

SUMMARY:
This study will be conducted to determine the effectiveness of education provided through the educational escape room method in nursing process teaching and to examine its effects on 4th-year nursing students' self-efficacy, teamwork, and anxiety.

DETAILED DESCRIPTION:
To improve and maintain the quality of nursing care, practices should be based on theoretical knowledge and carried out using the Nursing Process, which is a systematic scientific method. In line with the Nursing Process, the nurse plans, implements, and evaluates nursing interventions for the nursing diagnoses identified through the analysis and evaluation of the data collected regarding the health care needs of the healthy or ill individual. In addition to ensuring individualized and holistic care, the Nursing Process offers many benefits such as promoting critical thinking skills among nurses, enabling efficient use of time and energy in care delivery, distinguishing nursing practices from those of other health care professionals, and making nursing practice more visible. However, national and international studies emphasize that there are both individual and institutional barriers to the use of the Nursing Process in practice. In fact, related studies indicate that nurses experience difficulties in the diagnostic phase of the Nursing Process, particularly in making accurate nursing diagnoses and identifying etiological/related factors.

Therefore, it is important for nurses to acquire the necessary knowledge and skills for implementing nursing care in line with the Nursing Process during their nursing education. Nevertheless, studies have reported that students face challenges in understanding, planning, and applying the Nursing Process due to deficiencies in theoretical knowledge, practice, and experience, as well as inadequate problem-solving skills and difficulties in communication with health care professionals. In this context, it is recommended to incorporate active learning methods that complement traditional teaching methods in nursing education to ensure that nursing students understand and apply the importance of providing appropriate nursing care in accordance with the Nursing Process.

One of the active learning methods that has gained popularity in recent years is the educational escape room method. Educational escape rooms are designed to enable students to achieve specific learning outcomes by finding clues, solving puzzles, completing tasks within a limited time, and working collaboratively. The aim of this collaborative game is usually to escape from the room or to find a specific object. Escape rooms have been shown to significantly improve students' critical thinking and decision-making skills by encouraging them to analyze, evaluate, and solve problems, as well as contributing to the development of problem-solving skills and team collaboration. Among the skills that determine and strengthen problem-solving ability is self-efficacy; however, no study has been found that examines the effect of educational escape rooms on self-efficacy. Furthermore, the literature notes that the time limitation in this method may cause stress and anxiety among participants, yet some studies indicate that it can also reduce students' anxiety. Therefore, further research is needed to investigate the effects of educational escape rooms on self-efficacy and anxiety.

Although the literature on teaching the Nursing Process includes studies using active teaching methods such as virtual games, simulation, and web-based instruction, no study has been identified regarding the escape room method. It is believed that the use of the educational escape room method, an innovative active learning approach that complements traditional methods in teaching the Nursing Process, may be an effective strategy. Indeed, in line with the objectives of undergraduate education, nursing students are expected to graduate as professionals capable of implementing nursing care through the Nursing Process. In this regard, it is of critical importance to repeat interventions and trainings related to the teaching of the Nursing Process before students graduate. Within this scope, the present study will be conducted to determine the effectiveness of education provided through the educational escape room method in nursing process teaching and to examine its effects on 4th-year nursing students' self-efficacy, teamwork, and anxiety. This research will be conducted in a randomized experimental design with pretest-posttest experimental and control groups.The study sample will consist of senior nursing students who meet the inclusion criteria and agree to participate in the study. The students included in the sample will be randomly assigned to either the experimental or control group. The sample size of the study was calculated using a power analysis. Based on the data of a referenced study, the analysis indicated that with an effect size of 1.03, a power of 99%, and a significance level of 0.05 with a confidence interval, the required sample size was determined to be 62 fourth-year nursing students (a minimum of n=31 students per group). In order to increase the reliability of the study and to allow the use of parametric tests, the total sample size was determined as n=70, with 35 students in the experimental group and 35 students in the control group, taking into account possible data losses (such as dropouts). Randomization will be achieved through simple random sequencing using a randomization method. Participants will be randomly assigned to the experimental and control groups.Data will be analyzed using the SPSS (Statistical Package for Social Sciences) version 25.0 software. Data will be collected through the "Student Information Form," "Nursing Process Knowledge Test," "Self-Efficacy for Clinical Performance Scale," "Collaboration Scale," "State-Trait Anxiety Inventory," and the "Quality Measurement Tool for Nursing Diagnoses, Interventions, and Outcomes."

ELIGIBILITY:
Inclusion Criteria:

•Actively attending face-to-face education during the dates when the study will be conducted

Exclusion Criteria:

•Previous training with or familiarity with the educational escape room method

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-10-19 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Nursing Process Knowledge Test | 3 weeks before the intervention (before the theoretical nursing training) 2 weeks before the intervention (after the theoretical nursing process training) Directly after the intervention
  The form developed by the researcher in line with the literature regarding the stages of the Nursing Process consists of a total of 25 questions. Each correct answer is worth 4 points, with a maximum possible score of 100. The students' scores, whether low or high, will indicate their level of knowledge on the subject.
Skill in Applying the Nursing Care Plan | 1 week before the intervention (the first Nursing Process case study given after the theoretical nursing training) 2 weeks after the intervention (the second Nursing Process case study given after the intervention)
  To evaluate the quality and effectiveness of nursing process records, the "Quality Measurement Tool for Nursing Diagnoses, Interventions, and Outcomes" will be used. The scale consists of four sub-dimensions (Nursing Diagnoses as Process, Nursing Diagnoses as Outcomes, Nursing Interventions, and Nursing-Sensitive Patient Outcomes) and a total of 29 items. Higher scores on the scale indicate an increase in the quality of the nursing care plan.
Self-Efficacy | 3 weeks before the intervention 2 weeks after the intervention
  To determine nursing students' self-efficacy perceptions regarding clinical performance, the "Self-Efficacy Scale in Clinical Performance" will be used. The scale consists of a total of 37 items. It is a Likert-type scale with four sub-dimensions: data collection, diagnosis, implementation, and evaluation. The minimum possible mean item score is 0, and the maximum possible mean item score is 100. A higher score indicates a higher level of self-efficacy in clinical performance, while a lower score indicates a lower level of self-efficacy in clinical performance.
Team Collaboration | 3 weeks before the intervention Directly after the intervention
  To determine individuals' attitudes toward collaboration and their tendency to collaborate, the "Collaboration Scale" will be used. The scale consists of 11 items. It is a Likert-type scale with three sub-dimensions: emotions, behaviors, and beliefs. The minimum possible total score is 11 and the maximum is 55. Higher total scores on the scale indicate a higher tendency for collaboration.
Anxiety | 3 weeks before the intervention (Trait Anxiety Inventory) Directly before the intervention (State Anxiety Inventory) Directly after the intervention (State Anxiety Inventory)
  To determine individuals' anxiety levels, the State-Trait Anxiety Inventory (STAI) will be used. The scale consists of a total of 40 items and is a four-point Likert-type instrument composed of two subscales: the State Anxiety Inventory (first 20 items) and the Trait Anxiety Inventory (last 20 items). The State Anxiety subscale measures how an individual feels at a particular time and under specific conditions, whereas the Trait Anxiety subscale assesses how an individual generally feels regardless of the situation and conditions. A score between 0-19 indicates no anxiety, 20-39 indicates mild anxiety, 40-59 indicates moderate anxiety, and 60-79 indicates severe anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Aylin ÖZAKGÜL, Study Director — Istanbul University - Cerrahpasa
Locations (1):
- Bezmialem Vakif University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because the study is conducted as part of a doctoral thesis, and the collected data will be used only for the purposes of the study and related publications

REFERENCES:
- [Result] Chang YY, Chao LF, Xiao X, Chien NH. Effects of a simulation-based nursing process educational program: A mixed-methods study. Nurse Educ Pract. 2021 Oct;56:103188. doi: 10.1016/j.nepr.2021.103188. Epub 2021 Sep 3. PMID 34544010
- [Result] Ordu Y, Caliskan N. The effects of virtual gaming simulation on nursing students' diagnosis, goal setting, and diagnosis prioritization: A randomized controlled trial. Nurse Educ Pract. 2023 Mar;68:103593. doi: 10.1016/j.nepr.2023.103593. Epub 2023 Mar 2. PMID 36871387
- [Result] Chen D, Liu F, Zhu C, Tai C, Zhang Y, Wang X. The effect of an escape room game on college nursing students' learning attitude and game flow experiences in teaching safe medication care for the elderly: an intervention educational study. BMC Med Educ. 2023 Dec 12;23(1):945. doi: 10.1186/s12909-023-04961-3. PMID 38087301
- [Result] Molina-Torres G, Sandoval-Hernandez I, Ropero-Padilla C, Rodriguez-Arrastia M, Martinez-Cal J, Gonzalez-Sanchez M. Escape Room vs. Traditional Assessment in Physiotherapy Students' Anxiety, Stress and Gaming Experience: A Comparative Study. Int J Environ Res Public Health. 2021 Dec 3;18(23):12778. doi: 10.3390/ijerph182312778. PMID 34886502
- [Result] Rushdan EE, Mohamed MAE, Abdelhalim GE, El-Ashry AM, Ali HFM. Effect of an escape room as a gamification evaluation tool on clinical reasoning and teamwork skills among nursing students: A quasi-experimental study. Nurse Educ Pract. 2025 Jan;82:104188. doi: 10.1016/j.nepr.2024.104188. Epub 2024 Nov 14. PMID 39566365
- [Result] Quek LH, Tan AJQ, Sim MJJ, Ignacio J, Harder N, Lamb A, Chua WL, Lau ST, Liaw SY. Educational escape rooms for healthcare students: A systematic review. Nurse Educ Today. 2024 Jan;132:106004. doi: 10.1016/j.nedt.2023.106004. Epub 2023 Oct 24. PMID 37924674
- [Result] Gonzalez-de la Torre H, Hernandez-De Luis MN, Mies-Padilla S, Camacho-Bejarano R, Verdu-Soriano J, Rodriguez-Suarez CA. Effectiveness of "Escape Room" Educational Technology in Nurses' Education: A Systematic Review. Nurs Rep. 2024 May 13;14(2):1193-1211. doi: 10.3390/nursrep14020091. PMID 38804424
- [Result] Kalu F, Wolsey C, Enghiad P. Undergraduate nursing students' perceptions of active learning strategies: A focus group study. Nurse Educ Today. 2023 Dec;131:105986. doi: 10.1016/j.nedt.2023.105986. Epub 2023 Oct 17. PMID 37857101
- [Result] Rajabpoor, M., Zarifnejad, G. H., Mohsenizadeh, S. M., Mazloum, S. R., Pourghaznein, T., Mashmoul, A. & Mohammad, A. (2018). Barriers to the implementation of nursing process from the viewpoint of faculty members, nursing managers, nurses, and nursing students. Journal of Holistic Nursing and Midwifery, 28(2), 137-142.
- [Result] Rajabpoor M, Zarifnejad GH, Mohsenizadeh SM, Mazloum SR, Pourghaznein T, Mashmoul A, Mohammad A. Barriers to the implementation of nursing process from the viewpoint of faculty members, nursing managers, nurses, and nursing students. J Holist Nurs Midwifery. 2018;28(2):137-42.